CLINICAL TRIAL: NCT04010578
Title: Effects of Vitamin K2 and D3 Supplementation on 18F-NaF PET/MRI in Patients With Carotid and Coronary Artery Disease
Brief Title: Effects of VitamIN K2 and D3 supplementaTion on PET/MRI in Carotid Artery Disease
Acronym: INTRICATE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Academisch Ziekenhuis Maastricht (Other)
Collaborators: Horizon 2020 - European Commission (Other)
Responsible Party: Principal Investigator, Felix Mottaghy, Univ.-Prof. Dr. med., Academisch Ziekenhuis Maastricht
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL69450.068.19
Record Dates: First submitted 2019-07-01; First posted 2019-07-08 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Coronary Artery Disease; Carotid Artery Disease
Keywords: Vitamin K2; 18F-NaF; hybrid PET/MRI; Coronary artery calcification score; Menaquinone-7; Carotid Artery Disease; Coronary Artery Disease; Vitamin D3
MeSH Terms: conditions — Coronary Artery Disease; Carotid Artery Diseases | interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: One group will receive a MK-7 and vitamin D3 supplementation and the control group will receive a placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MK-7 and vitamin D3 supplementation (Experimental): Patients will receive a daily MK-7 and vitamin D3 supplementation for 3 months.
  Interventions: Dietary Supplement: MK-7 and vitamin D3
- Placebo (Placebo Comparator): Patients will receive a daily placebo for 3 months.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: MK-7 and vitamin D3 — Patients will receive 400 micro-grams of Menaquinone-7 and 80 micro-grams of vitamin D3 per day.
  Arms: MK-7 and vitamin D3 supplementation
Other: Placebo — Patients will receive a placebo each day.
  Arms: Placebo

SUMMARY:
Atherosclerosis is a disease of the arteries and is the result of various factors such as high blood cholesterol or diabetes, which lead to accumulations of fats, cells, and calcium deposits (i.e. plaques). It has been shown that people with a rapid increase in the amount of calcium deposits have a higher risk for stroke and heart attack than people with a decreased amount.

Previous scientific research has shown that a protein called Matrix Gla Protein plays an important role in the prevention of calcification. This protein works well only if there is enough Vitamin K in the blood vessels. In a large human studies, it has been shown that especially MK-7 (a form of Vitamin K2) is best absorbed by blood vessels. Moreover, studies suggest positive effects of vitamin D (especially D3) on vitamin K-dependent metabolism.

Over the last years, fluorine-18 sodium fluoride (18F-NaF) positron emission tomography (PET) emerged as a reliable clinical imaging tool able to detect micro-calcification in the blood vessels. Therefore, the present study will use 18F-NaF PET in combination with magnetic resonance imaging (MRI) to assess the influence of vitamin K and D supplementation in the development of arterial micro-calcification in the context of atherosclerosis.

The present study would like to confirm that MK-7 and vitamin D3 supplementation induces a significant reduction in the degree of micro-calcification from carotid artery disease patients, when comparing to a placebo, after 3 months.

This will be a prospective double blind randomised controlled feasibility study, in which one group will receive a MK-7 and vitamin D3 supplementation compared to a control group receiving a placebo.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic carotid artery disease on at least one side with a degree of stenosis > 25% (according to on the ECST criteria). If the patient has a symptomatic carotid artery disease on the contra-lateral side, he/she will still be included in the study, if intensified medical treatment for this symptomatic stenosis (e.g. statins, antiplatelet medication) was started ≥ 6 month before inclusion of the patient. This protocol was chosen in order to widely assure a stable situation on the plaque(s), which avoids an overspill from this medication on the assumed effects of the MK-7 and vitamin D3 supplementation.
* Age older than 18 years
* Signed informed consent provided

Exclusion Criteria:

* Antiplatelet or cholesterol lowering medication started within the past 6 months
* Chronic or paroxysmal atrial fibrillation
* Presence or scheduled coronary or carotid revascularisation procedure (e.g. stent implantation, coronary artery bypass graft, balloon-dilatation, endarterectomy, angioplasty)
* History of myocardial infarction or stroke
* Malignant disease (except for treated basal-cell or squamous cell carcinoma)
* Use of vitamin K antagonists or any other anticoagulation treatment
* A life-expectancy < 1 year
* Claustrophobia
* Presence of a pacemaker, intra-cardiac defibrillator, or metallic implant (e.g. vascular clip, neuro-stimulator, cochlear implant)
* Body weight > 130kg or body habitus that does not fit into the gantry
* Pregnancy or wish to become pregnant in the near future
* Breast feeding
* (History of) metabolic or gastrointestinal disease
* Use of vitamin K or D containing supplements or vitamin K-rich foods (i.e. soya)
* Chronic inflammatory disease
* Systemic treatment or topical treatment likely to interfere with evaluation of the study parameters
* Corticoid treatment
* Participation in a clinical study more recently than one month before the current study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
The change in time of vascular micro-calcification via (18)F-NaF PET/MRI | 3 months follow-up
  The primary outcome of this study is the mean rate of the change in time of vascular micro-calcification in the carotid arteries, measured as a difference between the intervention group and placebo group in (18)F-NaF uptake via hybrid PET/MRI after the 3 months of treatment.

SECONDARY OUTCOMES:
The change in time of vascular calcification via coronary artery calcification score | 3 months follow-up
  Investigating whether MK-7 and vitamin D3 supplementation can diminish, halt or even reverse the development of arterial micro-calcification in the coronary arteries, measured as a difference between the intervention group and placebo group in coronary artery calcification score after the 3 months.
  The Agatston coronary artery calcification score isis a semi-automated tool to calculate a score based on the extent of coronary artery calcification detected by an non-contrast low-dose CT scan. The score ranges from 0 arbitrary units to > 400. The higher the value of the score, the higher the degree of calcification is in the coronary arteries; hence, lower values usually represent a better outcome.
The correlation between (18)F-NaF PET/MRI and coronary artery calcification score | 3 months follow-up
  The correlation between the uptake of (18)F-NaF at 3 months and the coronary artery calcification score.
  The Agatston coronary artery calcification score isis a semi-automated tool to calculate a score based on the extent of coronary artery calcification detected by an non-contrast low-dose CT scan. The score ranges from 0 arbitrary units to > 400. The higher the value of the score, the higher the degree of calcification is in the coronary arteries; hence, lower values usually represent a better outcome.
The influence of MK-7 and vitamin D3 supplementation on MRI parameters | baseline vs 3 months follow-up
  Investigating whether MK-7 and vitamin D3 supplementation can influence the fibrous cap status on the MRI.

OTHER OUTCOMES:
The influence of MK-7 and vitamin D3 supplementation on carotid intima-media thickness | baseline vs 3 months follow-up
  Investigating whether MK-7 and vitamin D3 supplementation can influence the carotid intima-media thickness

CONTACTS AND LOCATIONS:
Overall Officials: Felix M Mottaghy, MD, PhD, Principal Investigator — Maastricht University Medical Center

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be shared.
Supporting Information: SAP, ICF
Time Frame: IPD will be shared stating with 6 months after publication.
Access Criteria: Access criteria will be discussed with all the study members, then it will be published.